CLINICAL TRIAL: NCT05667558
Title: Assessment of Intake of Energy and Selected Nutrients, Nutritional Status, Body Composition and Biochemical Parameters of Obese Patients Before and After Bariatric Surgery
Brief Title: Assessment of the Clinical Condition and Way of Nutrition Patients Before and After Sleeve Gastrectomy
Status: Completed | Type: Observational
Sponsor: Medical University of Bialystok (Other)
Responsible Party: Sponsor
Other Study IDs: N/ST/MN/18/001/3316
Record Dates: First submitted 2022-12-01; First posted 2022-12-28 (Actual); Last update posted 2022-12-28 (Actual); Status verified 2022-11

CONDITIONS: Obesity
Keywords: bariatric surgery; nutrition; body composition; nutritional status; obesity; laparoscopic sleeve gastrectomy
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study grup

SUMMARY:
Conservative treatment of patients with morbid obesity is inefficient, which is why surgical treatment is necessary. Although bariatric treatment is associated with the occurrence of complications resulting from the procedure or from nutritional insufficiencies, it leads to significant body mass reduction and metabolic improvement of obese patients.

The aim of the study was to determine the clinical condition of obese patients after laparoscopic sleeve gastrectomy ( LSG) in terms of nutritional status, metabolic disorders and way of nutrition.

The study conduced 4 visits: preliminary visit (1 day before the surgery) and control visits (1, 3 and 6 months after the surgery). Based on the inclusion and exclusion criteria the observational study was conducted among 30 participants (15 women and 15 men).

ELIGIBILITY:
Inclusion criteria

* women and men aged 18-64
* BMI ≥ 40 kg/m2 or BMI ≥ 35 kg/m2 with comorbidities such as type II diabetes (T2DM), hypertension, sleep apnea and other respiratory disorders, non-alcoholic fatty liver disease, osteoarthritis, lipid abnormalities, gastrointestinal disorders, or heart disease

Exclusion Criteria:

* pregnancy
* gastrointestinal cancers
* cardiorespiratory failure

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study included 30 obese patients (15 women and 15 man) who met the criteria for beaing included in the study and who did not possess excusion criteria.inclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2017-11-30 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Changes in anthropometric measurements during the 6 months after surgery | before and 1,3 and 6 months after LSG
  Body weight in kilograms was measured using a scale with stadiometer. Body height in meters was measured using a scale with stadiometer. Body weight and height were used to calculate BMI (Body Mass Index) in kilograms divided by square metres.
  Hip circumference in centimeters was measured at the greater trochanters at the widest part of the hips. Waist circumference in centimeters was measured at the uppermost lateral border of the hip crest.
Changes in percentage of excess weight loss during the 6 months after surgery | 1, 3 and 6 months after LSG
  Percentage of excess weight loss (%EWL) was calculated using the formula:
  %EWL = (preoperative weight - current weight)/(preoperative weight - ideal weight) × 100.
  Ideal body weight was calculated using Lorentz formula.
Changes in body composition during the 6 months after surgery | before and 1,3 and 6 months after LSG
  Body composition was assessed four times (before and 1,3 and 6 months after LSG). Body composition parameters (fat mass in kilograms, percentage of body fat, fat free mass in kilograms, percentage of fat free mass, total body water in liters, percentage of total body water) was determined using the bioelectrical impedance method (BioScan 920-2 body composition analyzer, Maltron International Ltd., United Kingdom)
Changes in energy and selected nutrients intake during the 6 months after surgery | before and 1,3 and 6 months after LSG
  The intake of energy and selected nutrients was assessed four times (before and 1,3 and 6 months after LSG). A 3-day nutrition interview was collected. The supply of energy, protein, fat (including fatty acids), carbohydrates, dietary fibre, vitamins and minerals in the usual diet was assessed.
Changes in blood biochemical parameters of patients during the 6 months after surgery. | before and 1,3 and 6 months after LSG
  The biochemical parameters of the patient's blood were assessed four times (before and 1,3 and 6 months after LSG). Laboratory tests were performer to determine the following serum levels: fasting glucose, fasting insulin,total cholesterol, LDL cholesterol fraction, HDL cholesterol fraction, triglycerides and aminotransferases: alanine (ALT) and aspartate (AST), complete blood count.
  The HOMA-IR (homeostasis model assessment of insulin resistance) index was calculated according to the formula: [fasting insulin (mIU/l) x fasting glucose (mg/dl)] / 405

CONTACTS AND LOCATIONS:
Overall Officials: Lucyna Ostrowska, Professor, Study Director — Department of Dietetics and Clinical Nutrition Medical University of Bialystok
Locations (1):
- Medical University of Bialystok, Bialystok, Poland

REFERENCES:
- [Background] Chang SH, Stoll CR, Song J, Varela JE, Eagon CJ, Colditz GA. The effectiveness and risks of bariatric surgery: an updated systematic review and meta-analysis, 2003-2012. JAMA Surg. 2014 Mar;149(3):275-87. doi: 10.1001/jamasurg.2013.3654. PMID 24352617
- [Background] Al-Mutawa A, Anderson AK, Alsabah S, Al-Mutawa M. Nutritional Status of Bariatric Surgery Candidates. Nutrients. 2018 Jan 11;10(1):67. doi: 10.3390/nu10010067. PMID 29324643
- [Background] Sherf Dagan S, Zelber-Sagi S, Webb M, Keidar A, Raziel A, Sakran N, Goitein D, Shibolet O. Nutritional Status Prior to Laparoscopic Sleeve Gastrectomy Surgery. Obes Surg. 2016 Sep;26(9):2119-2126. doi: 10.1007/s11695-016-2064-9. PMID 26797718
- [Background] Batar N, Pulat Demir H, Bayram HM. Assessment of nutritional status, body composition and blood biochemical parameters of patients following sleeve gastrectomy: 6 months follow up. Clin Nutr ESPEN. 2021 Jun;43:184-190. doi: 10.1016/j.clnesp.2021.04.016. Epub 2021 Apr 27. PMID 34024512
- [Background] Sherf Dagan S, Tovim TB, Keidar A, Raziel A, Shibolet O, Zelber-Sagi S. Inadequate protein intake after laparoscopic sleeve gastrectomy surgery is associated with a greater fat free mass loss. Surg Obes Relat Dis. 2017 Jan;13(1):101-109. doi: 10.1016/j.soard.2016.05.026. Epub 2016 Jun 2. PMID 27521254
- [Background] Dulloo AG, Jacquet J, Miles-Chan JL, Schutz Y. Passive and active roles of fat-free mass in the control of energy intake and body composition regulation. Eur J Clin Nutr. 2017 Mar;71(3):353-357. doi: 10.1038/ejcn.2016.256. Epub 2016 Dec 14. PMID 27966570
- [Background] Friedrich AE, Damms-Machado A, Meile T, Scheuing N, Stingel K, Basrai M, Kuper MA, Kramer KM, Konigsrainer A, Bischoff SC. Laparoscopic sleeve gastrectomy compared to a multidisciplinary weight loss program for obesity--effects on body composition and protein status. Obes Surg. 2013 Dec;23(12):1957-65. doi: 10.1007/s11695-013-1036-6. PMID 23856991
- [Background] Hopkins M, Finlayson G, Duarte C, Whybrow S, Ritz P, Horgan GW, Blundell JE, Stubbs RJ. Modelling the associations between fat-free mass, resting metabolic rate and energy intake in the context of total energy balance. Int J Obes (Lond). 2016 Feb;40(2):312-8. doi: 10.1038/ijo.2015.155. Epub 2015 Aug 17. PMID 26278004
- [Background] Fuchs T, Loureiro M, Both GH, Skraba HH, Costa-Casagrande TA. THE ROLE OF THE SLEEVE GASTRECTOMY AND THE MANAGEMENT OF TYPE 2 DIABETES. Arq Bras Cir Dig. 2017 Oct-Dec;30(4):283-286. doi: 10.1590/0102-6720201700040013. PMID 29340555
- [Background] Yip S, Plank LD, Murphy R. Gastric bypass and sleeve gastrectomy for type 2 diabetes: a systematic review and meta-analysis of outcomes. Obes Surg. 2013 Dec;23(12):1994-2003. doi: 10.1007/s11695-013-1030-z. PMID 23955521
- [Background] Milone M, Lupoli R, Maietta P, Di Minno A, Bianco P, Ambrosino P, Coretti G, Milone F, Di Minno MN, Musella M. Lipid profile changes in patients undergoing bariatric surgery: a comparative study between sleeve gastrectomy and mini-gastric bypass. Int J Surg. 2015 Feb;14:28-32. doi: 10.1016/j.ijsu.2014.12.025. Epub 2015 Jan 7. PMID 25576760
- [Background] Bower G, Toma T, Harling L, Jiao LR, Efthimiou E, Darzi A, Athanasiou T, Ashrafian H. Bariatric Surgery and Non-Alcoholic Fatty Liver Disease: a Systematic Review of Liver Biochemistry and Histology. Obes Surg. 2015 Dec;25(12):2280-9. doi: 10.1007/s11695-015-1691-x. PMID 25917981